CLINICAL TRIAL: NCT05575817
Title: Web Based Therapist and Patient Tutorials on Prolonged Grief. Study 2
Brief Title: Web Based Patient Tutorial on Prolonged Grief
Acronym: STTR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Center for Psychological Consultation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Shear, MD, Marion E. Kenworthy Professor of Psychiatry, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAT7389 Study2; 1R41MH118126-01A1 (NIH)
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Prolonged Grief Disorder
Keywords: grief; therapy; training
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: Study 2 is an open-label (non-randomized) pilot study to determine therapist and patient acceptance, feasibility and whether there is enough of a signal in improving clinical outcomes to warrant a randomized trial of the online patient grief tutorial in conjunction with Prolonged Grief Disorder therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient online grief tutorial (Experimental): Participants will be given access to an online 9-module interactive tutorial about grief to be used in conjunction with a course of Prolonged Grief Disorder Therapy.
  Interventions: Behavioral: Web Based Patient Tutorial on Prolonged Grief Disorder Therapy

INTERVENTIONS:
Behavioral: Web Based Patient Tutorial on Prolonged Grief Disorder Therapy — The patient tutorial will contain 9 modules, each designed to be used flexibly in conjunction with Prolonged Grief Disorder Therapy (PGDT) telehealth sessions with the therapist. Each module takes about 15-30 minutes to complete. The patient tutorial consists of information about grief and adaptation to loss, including a description of seven healing milestones that are the focus of PGDT and an explanation of prolonged grief and how to understand it. In addition, the tutorial has descriptions of the procedure, goals and rationale for a series of in-session therapeutic exercises to be undertaken with the therapist, as well as descriptions and encouragement to participate in interim therapeutic activities (i.e., "homework") assigned by the therapist after each treatment session. The tutorial also contains a self-assessment component for each module that can be completed by the patient and shared with the therapist.

SUMMARY:
The goal of this clinical trial is to learn about usefulness of the online patient grief tutorial in bereaved adults with Prolonged Grief Disorder who are receiving psychotherapy treatment for it. The main question it aims to answer is how helpful the tutorial was and how much therapists and clients liked it.

Participants will be given access to the online tutorial for use during their talk therapy treatment. Participants will be asked to complete surveys before starting the treatment and after its completion to provide information about their symptoms and feedback about the tutorial.

DETAILED DESCRIPTION:
The Center for Prolonged Grief at Columbia University will send announcements to therapists who have done training in Prolonged Grief Disorder Treatment (PGDT) inviting them to participate in the study and directing them to a study information page in Qualtrics. After reviewing the information sheet, therapists will give their consent for participation and then complete a demographics and professional experience questionnaire. The study coordinator will monitor Qualtrics for new responses and email eligible therapist-participants instructions for accessing the tutorial in Moodle.

Participating therapists will then recruit their patients to take part in the study and direct them to the study information page in Qualtrics to provide consent. Therapists will conduct a clinical assessment to determine that the client is an appropriate candidate for the study. Then therapists will provide the clients with a brief introduction to the patient tutorial and log-in credentials, before starting Prolonged Grief Disorder Treatment. Client-participants will have access to the tutorial for 6 months.

The patient tutorial will supplement a course of Prolonged Grief Disorder Treatment (aka Complicated Grief Treatment or CGT) provided by participating therapists in their practices. Typical course of PGDT takes about 4 months of weekly meetings. Therapists are licensed professionals who will monitor their patients, as usual in practice, and can recommend to stop the study treatment at any point or switch to alternative treatment, as indicated. Frequency, duration and pattern of use of the patient online tutorial will be monitored. Patients will also complete online questionnaires about their grief symptoms before and after treatment and overall experience with the tutorial.

ELIGIBILITY:
Licensed mental health professionals trained in prolonged grief disorder treatment and their clients in treatment for prolonged grief.

Inclusion criteria to participate in step 2 of the study are:

1. a clinical diagnosis of prolonged grief disorder according to DSM-5 criteria,
2. a judgment that grief is the primary problem,
3. a score of at least 30 on the Inventory for Complicated Grief (ICG), and
4. at least 1 year has passed after the death of their loved one (part of DSM-5 criteria).

Exclusion criteria:

1) active suicidal ideation or suicidal intent, current or past psychotic disorder, or active substance use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Patient feedback survey | Up to 6 months (treatment completion)
  This is a 7-item questionnaire about usefulness of the tutorial; 4 items are rated from 1 (strongly disagree) to 5 (strongly agree) and are added for a composite total score (range 4-20) with higher scores indicating greater usefulness (better outcome). 3 remaining items solicit open-ended written feedback.
Therapist feedback survey | Up to 6 months (treatment completion)
  This is a 6-item questionnaire about usefulness of the tutorial where 3 items are rated from 1 (strongly disagree) to 5 (strongly agree)and are added for a composite total score (range 3-15) with higher scores indicating greater usefulness (better outcome). 3 remaining items solicit open-ended written feedback.

SECONDARY OUTCOMES:
Inventory of Complicated Grief | Change from baseline to 6 months (before and after treatment completion)
  This is a 19-item questionnaire assessing prolonged grief symptoms. Each item is rated on a scale 0-4 to produce a total score ranges from 0 to 76, with higher scores indicating more severe grief (worse outcome).
Work and Social Adjustment Scale | Change from baseline to 6 months (before and after treatment completion)
  This is a self-report scale assessing grief interference in 5 areas of functioning, rated 0-8, with a total score ranging from 0 to 40 with higher scores indicating more interference (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Kobak, PhD, Principal Investigator — Center for Psychological Consulation; Katherine Shear, MD, Principal Investigator — Columbia School of Social Work
Locations (2):
- United States (2):
  - Center for Complicated Grief, Columbia School of Social Work, New York, New York
  - Center for Psychological Consultation, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Background] Shear MK, Reynolds CF 3rd, Simon NM, Zisook S, Wang Y, Mauro C, Duan N, Lebowitz B, Skritskaya N. Optimizing Treatment of Complicated Grief: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jul 1;73(7):685-94. doi: 10.1001/jamapsychiatry.2016.0892. PMID 27276373